CLINICAL TRIAL: NCT05023031
Title: A Phase 1 Clinical Trial, Open-label, Randomized Study in Healthy Subjects to Evaluate Pharmacokinetic Characteristics and Safety After Oral Administration of NVP-2102 and NVP-2102-R in Healthy Subjects
Brief Title: Evaluation of Pharmacokinetic and Safety of NVP-2102 and NVP-2102-R in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-2102_BE
Record Dates: First submitted 2021-07-05; First posted 2021-08-26 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-2102 (Experimental): NVP-2102
  Interventions: Drug: NVP-2102
- NVP-2102-R (Active Comparator): NVP-2102-R
  Interventions: Drug: NVP-2102-R

INTERVENTIONS:
Drug: NVP-2102 — Tablet formulation for oral administration, single dose of NVP-2102 at Day 1
  Arms: NVP-2102
Drug: NVP-2102-R — Tablet formulation for oral administration, single dose of NVP-2102-R at Day 1
  Arms: NVP-2102-R

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety of NVP-2102 and NVP-2102-R.

DETAILED DESCRIPTION:
Evaluate the pharmacokinetics and safety of NVP-2102 compared to NVP-2102-R

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject, 19 years of age or older
* Subjects who signed informed consent
* Body mass index(BMI) of 18 to 30.0 kg/㎡

Exclusion Criteria:

* Subject who has clinically significant medical history
* Inadequate subject for the clinical trial by the investigator's decision
* Subjects participated in another clinical trial within 6 months prior to the first administration of investigational product

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Area under the plasma drug concentration-time curve(AUCt) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Maximum observed plasma concentration(Cmax) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma

SECONDARY OUTCOMES:
Evaluation of Area under the plasma drug concentration-time curve from time 0 to infinity(AUC∞) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of AUCt/AUC∞ | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Time of peak concentration(Tmax) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of Terminal phase of Half-life(t1/2) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of total clearance of the drug from plasma after oral administration(CL/F) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma
Evaluation of volume of distribution after non-intravenous administration(Vz/F) | 0 ~ 72 hours
  Pharmacokinetics parameter derived from plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jae Woo Kim, Principal Investigator — H+ Yangji hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Nambusunhwan-ro, South Korea

IPD SHARING:
Plan to Share IPD: No